CLINICAL TRIAL: NCT04535401
Title: Phase I/Ib Trial of ATR Inhibitor BAY 1895344 in Combination With FOLFIRI in GI Malignancies With a Focus on Metastatic Colorectal and Gastric/Gastroesophageal Cancers
Brief Title: Testing the Addition of an Anticancer Drug, BAY 1895344, to the Usual Chemotherapy With FOLFIRI in Advanced or Metastatic Cancers of the Stomach and Intestines
Status: Active, not recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: NCI-2020-06482; NCI-2020-06482 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); 21-060; 10406 (Other: UPMC Hillman Cancer Center LAO); 10406 (Other: CTEP); UM1CA186690 (NIH)
Record Dates: First submitted 2020-09-01; First posted 2020-09-02 (Actual); Last update posted 2024-10-10 (Actual); Status verified 2024-04

CONDITIONS: Advanced Colorectal Carcinoma; Advanced Digestive System Carcinoma; Advanced Gastric Carcinoma; Advanced Gastroesophageal Junction Adenocarcinoma; Clinical Stage III Gastric Cancer AJCC v8; Clinical Stage III Gastroesophageal Junction Adenocarcinoma AJCC v8; Clinical Stage IV Gastric Cancer AJCC v8; Clinical Stage IV Gastroesophageal Junction Adenocarcinoma AJCC v8; Metastatic Colorectal Carcinoma; Metastatic Digestive System Carcinoma; Metastatic Gastric Carcinoma; Metastatic Gastroesophageal Junction Adenocarcinoma; Stage III Colorectal Cancer AJCC v8; Stage IV Colorectal Cancer AJCC v8
MeSH Terms: conditions — Colorectal Neoplasms; Stomach Neoplasms | interventions — Biopsy; Specimen Handling; X-Rays; BAY 1895344; Fluorouracil; dehydroftorafur; Irinotecan; Leucovorin

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Treatment (elimusertib, FOLFIRI) (Experimental): Patients receive elimusertib PO QD on days 2, 3, 16, and 17 and irinotecan hydrochloride IV over 90 minutes, fluorouracil IV over 46 hours, and leucovorin calcium IV on days 1 and 15. Cycles repeat every 28 day in the absence of disease progression or unacceptable toxicity. Patients undergo tumor biopsy during screening and on study and blood sample collection and imaging throughout the study.
  Interventions: Procedure: Biopsy; Procedure: Biospecimen Collection; Procedure: Diagnostic Imaging; Drug: Elimusertib; Drug: Fluorouracil; Drug: Irinotecan Hydrochloride; Drug: Leucovorin Calcium

INTERVENTIONS:
Procedure: Biopsy — Undergo tumor biopsy
  Other Names: BIOPSY_TYPE; Bx
Procedure: Biospecimen Collection — Undergo blood sample collection
  Other Names: Biological Sample Collection; Biospecimen Collected; Specimen Collection
Procedure: Diagnostic Imaging — Undergo imaging
  Other Names: Medical Imaging
Drug: Elimusertib — Given PO
  Other Names: ATR Inhibitor BAY1895344; ATR Kinase Inhibitor BAY1895344; BAY 1895344; BAY-1895344; BAY1895344
Drug: Fluorouracil — Given IV
  Other Names: 5 Fluorouracil; 5 Fluorouracilum; 5 FU; 5-Fluoro-2,4(1H, 3H)-pyrimidinedione; 5-Fluorouracil; 5-Fluracil; 5-Fu; 5FU; AccuSite; Carac; Fluoro Uracil; Fluouracil; Flurablastin; Fluracedyl; Fluracil; Fluril; Fluroblastin; Ribofluor; Ro 2-9757; Ro-2-9757
Drug: Irinotecan Hydrochloride — Given IV
  Other Names: Campto; Camptosar; Camptothecin 11; Camptothecin-11; CPT 11; CPT-11; CPT11; Irinomedac; Irinotecan Hydrochloride Trihydrate; Irinotecan Monohydrochloride Trihydrate; U 101440E; U-101440E; U101440E
Drug: Leucovorin Calcium — Given IV
  Other Names: Adinepar; Calcifolin; Calcium (6S)-Folinate; Calcium Folinate; Calcium Leucovorin; Calfolex; Calinat; Cehafolin; Citofolin; Citrec; Citrovorum Factor; Cromatonbic Folinico; Dalisol; Disintox; Divical; Ecofol; Emovis; Factor, Citrovorum; Flynoken A; Folaren; Folaxin; FOLI-cell; Foliben; Folidan; Folidar; Folinac; Folinate Calcium; folinic acid; Folinic Acid Calcium Salt Pentahydrate; Folinoral; Folinvit; Foliplus; Folix; Imo; Lederfolat; Lederfolin; Leucosar; leucovorin; Rescufolin; Rescuvolin; Tonofolin; Wellcovorin

SUMMARY:
This phase I trial investigates the best dose, possible benefits and/or side effects of BAY 1895344 in combination with FOLFIRI in treating patients with stomach or intestinal cancer that that may have spread from where it first started to nearby tissue, lymph nodes, or distant parts of the body (advanced) or has spread from where it first started (primary site) to other places in the body (metastatic). BAY 1895344 may stop the growth of tumor cells by blocking some of the enzymes needed for cell growth. Chemotherapy drugs, such as irinotecan, fluorouracil, and leucovorin, (called FOLFIRI in short) work in different ways to stop the growth of tumor cells, either by killing the cells, by stopping them from dividing, or by stopping them from spreading. Giving BAY 1895344 in combination with FOLFIRI may help shrink advanced or metastatic stomach and/or intestinal cancer.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVE:

I. Determine the safety and maximum tolerated dose (MTD) of elimusertib (BAY 1895344) with leucovorin calcium, fluorouracil, and irinotecan hydrochloride (FOLFIRI).

SECONDARY OBJECTIVES:

I. To observe and record anti-tumor activity by overall response rate (ORR), progression-free survival (PFS), and overall survival (OS).

II. Determine the response and clinical benefit rate (complete response + partial response + stable disease) of BAY 1895344 with FOLFIRI in colorectal and gastric/gastroesophageal cancers.

III. Evaluate tumor and peripheral blood mononuclear cell (PBMC) deoxyribonucleic acid (DNA) damage signaling in the context of the chemotherapy backbone alone and when combined with BAY 1895344.

IV. Evaluate the pharmacokinetics (PK) profile of fluorouracil (5-FU) and irinotecan.

V. Evaluate the PK profile of BAY 1895344. VI. Evaluate the relationship between ATM status by immunohistochemistry (IHC) and clinical efficacy of the BAY 1895344/FOLFIRI combination.

EXPLORATORY OBJECTIVES:

I. Evaluate the exposure-response relationship between drug exposures and toxicity and response, and UGT1A1 genotype.

II. Evaluate the relationship between tumor mutations and clinical efficacy of the BAY 1895344/FOLFIRI combination.

OUTLINE: This is a dose-escalation study of elimusertib, irinotecan, and fluorouracil with fixed-dose leucovorin followed by a dose-expansion study.

Patients receive elimusertib orally (PO) once daily (QD) on days 2, 3, 16, and 17 and irinotecan hydrochloride intravenously (IV) over 90 minutes, fluorouracil IV over 46 hours, and leucovorin calcium IV on days 1 and 15. Cycles repeat every 28 day in the absence of disease progression or unacceptable toxicity. Patients undergo tumor biopsy during screening and on study and blood sample collection and imaging throughout the study.

After completion of study treatment, patients are followed up for 30 days and then every 3 months for up to 1 year or until their disease gets worse or they begin a new treatment for their cancer.

ELIGIBILITY:
Inclusion Criteria:

* For Dose Escalation: Patients must have histologically or cytologically confirmed advanced or metastatic gastrointestinal (GI) cancers with Response Evaluation Criteria in Solid Tumors 1.1 (RECIST1.1) measurable disease who have progressed on at least one prior treatment for metastatic disease and for whom FOLFIRI is considered a reasonable treatment option. Patients with mismatch repair deficiency should have progressed on immunotherapy
* For Dose Expansion: Patients must have either:

  * Colorectal cancer who have previously progressed on irinotecan and tolerated an irinotecan dose equal to or greater than the recommended phase 2 dose (RP2D). If they have mismatch repair deficiency they should have progressed on immunotherapy OR
  * Gastroesophageal cancer who have progressed on at least one first-line therapy for metastatic disease. If they have mismatch repair deficiency they should have progressed on immunotherapy
* For Dose Expansion: Patients be willing to undergo biopsies for research purposes only. The accessible tumor can be the primary or metastatic tumor site. Both research biopsies should be taken from the same tumor site
* Patients must have progressive disease on at least first-line therapy for metastatic disease. Previous treatment with irinotecan is allowed
* Age >= 18 years. Because no dosing or adverse event data are currently available on the use of BAY 1895344 in combination with FOLFIRI in patients <18 years of age, children are excluded from this study
* Eastern Cooperative Oncology Group (ECOG) performance status =< 1
* Leukocytes >= 3,000/mcL
* Absolute neutrophil count >= 1,500/mcL
* Platelets >= 100,000/mcL
* Total bilirubin =< 1.5 x institutional upper limit of normal (ULN)
* Aspartate aminotransferase (AST) (serum glutamic-oxaloacetic transaminase [SGOT])/alanine aminotransferase (ALT) (serum glutamate pyruvate transaminase [SGPT]) =< 3 x institutional ULN
* Glomerular filtration rate (GFR) >= 60 mL/min/1.73 m^2 using the Chronic Kidney Disease Epidemiology Collaboration (CKD-EPI) equation
* International normalization ratio (INR) =< 1.5 × ULN unless participant is receiving anticoagulant therapy, in which case prothrombin time (PT) or activated partial thromboplastin time (aPTT) should be within expected therapeutic range of anticoagulants. If patient has a new diagnosis of venous thromboembolism (VTE), then patient should be appropriately anticoagulated with low molecular weight heparin (LMWH) or direct acting oral anticoagulants (DOACs) and be clinically stable for at least 1 week post treatment onset
* Human immunodeficiency virus (HIV)-infected patients on effective anti-retroviral therapy, that does not interact with study therapy, with undetectable viral load within 6 months are eligible for this trial
* For patients with evidence of chronic hepatitis B virus (HBV) infection, the HBV viral load must be undetectable on suppressive therapy that does not interact with study therapy, if indicated
* Patients with a history of hepatitis C virus (HCV) infection must have been treated and cured. For patients with HCV infection who are currently on treatment, they are eligible if they have an undetectable HCV viral load and HCV therapy does not interact with study therapy
* Patients with treated brain metastases are eligible if follow-up brain imaging after central nervous system (CNS)-directed therapy shows no evidence of progression
* Patients with a prior or concurrent malignancy whose natural history or treatment does not have the potential to interfere with the safety or efficacy assessment of the investigational regimen are eligible for this trial
* Patients with known history or current symptoms of cardiac disease, or history of treatment with cardiotoxic agents, should have a clinical risk assessment of cardiac function using the New York Heart Association Functional Classification. To be eligible for this trial, patients should be class 2B or better
* The effects of BAY 1895344 on the developing human fetus are unknown. For this reason and because DNA-damage response inhibitors agents as well as other therapeutic agents used in this trial, 5-FU and irinotecan, are known to be teratogenic, women of child-bearing potential and men must agree to use adequate contraception (hormonal or barrier method of birth control; abstinence) prior to study entry and for the duration of study participation and for 6 months after completion of BAY 1895344 administration

  * Should a woman become pregnant or suspect she is pregnant while she or her partner is participating in this study, she should inform her treating physician immediately. Men treated or enrolled on this protocol must also agree to use adequate contraception prior to the study, for the duration of study participation, and 6 months after completion of study treatment administration
* Ability to understand and the willingness to sign a written informed consent document. Participants with impaired decision-making capacity (IDMC) who have a legally-authorized representative (LAR) and/or family member available will also be eligible

Exclusion Criteria:

* Patients with a history of prior treatment with an ATR inhibitor
* Patients with a history of other malignancy that could affect compliance with the protocol or interpretation of the results
* Patients who have had chemotherapy or radiotherapy within 3 weeks (6 weeks for nitrosoureas or mitomycin C) prior to entering the study
* Patients who have not recovered from adverse events due to prior anti-cancer therapy (i.e., have residual toxicities > grade 1) with the exception of alopecia
* Patients who are receiving any other investigational agents
* History of hypersensitivity or allergic reactions attributed to compounds of similar chemical or biologic composition to BAY 1895344, 5-FU, leucovorin, or irinotecan. Patient eligibility can be discussed with the primary investigator (PI) if prior reactions do not seem to warrant excluding the patient
* Patients receiving any medications that are substrates of CYP3A4 with a narrow therapeutic window or strong inhibitors/inducers of CYP3A4 are ineligible, if they cannot be transferred to alternative medication. Because the lists of these agents are constantly changing, it is important to regularly consult a frequently-updated medical reference. As part of the enrollment/informed consent procedures, the patient will be counseled on the risk of interactions with other agents, and what to do if new medications need to be prescribed or if the patient is considering a new over-the-counter medicine or herbal product
* Patients with uncontrolled intercurrent illness
* Patients with psychiatric illness/social situations that would limit compliance with study requirements
* Gastrointestinal pathology or history that adversely impact the ability to take or absorb oral medication
* Pregnant women are excluded from this study because BAY 1895344 as a DNA-damage response inhibitor may have the potential for teratogenic or abortifacient effects. Because there is an unknown but potential risk for adverse events in nursing infants secondary to treatment of the mother with BAY 1895344 breastfeeding should be discontinued if the mother is treated with BAY 1895344 and for 4 months after end of treatment. These potential risks may also apply to other agents used in this study
* Patients who were unable to tolerate prior irinotecan treatment are excluded from this study
* Patients with a corrected QT (QTc) interval >= 470 msec are excluded from this study

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 10 (Actual)
Dates: Start 2021-08-13 (Actual); Primary Completion 2024-03-29 (Actual); Study Completion 2025-04-29 (Estimated)

PRIMARY OUTCOMES:
Maximum tolerated dose (MTD) of elimusertib (BAY 1895344) in combination with irinotecan, fluorouracil, and leucovorin (FOLFIRI) | Up to 28 days
  A BOIN - Bayesian Optimal intervals trial design will be used to determine the MTD.

SECONDARY OUTCOMES:
Overall response rate | Up to 1 year post treatment
  Assessed per Response Evaluation Criteria in Solid Tumors. The probability of clinical response (complete response [CR]+partial response [PR]) and disease control (CR+PR+stable disease) will be estimated within the disease cohorts, with consideration of previous irinotecan exposure, with exact 95% binomial confidence intervals.
Progression-free survival (PFS) | From start of treatment to time of progression or death, whichever occurs first, assessed up to 1 year
  PFS will be estimated within disease cohorts by the product-limit (Kaplan-Meier) estimator, along with 95% confidence regions.
Overall survival (OS) | Up to 1 year post treatment
  OS will be estimated within disease cohorts by the product-limit (Kaplan-Meier) estimator, along with 95% confidence regions.
Peripheral blood mononuclear cell gammaH2AX and p-ATM signaling | Up to 1 year post treatment
  Signaling during the pharmacokinetics (PK) lead-in and in combination with BAY 1895344 will be compared with a non-parametric paired test (e.g. Wilcoxon rank test), at a significance level at p < 0.05. For tumors, this will be performed only for patients in the dose expansion cohorts.
Tumor multiplex immunofluorescence assay signaling | Up to 1 year post treatment
  Signaling during the PK lead-in and in combination with BAY 1895344 will be compared with a non-parametric paired test (e.g. Wilcoxon rank test), at a significance level at p < 0.05. For tumors, this will be performed only for patients in the dose expansion cohorts.
Area under curve (AUC) and concentration maximum (Cmax) of irinotecan and 5-FU | Up to 1 year post treatment
  PK during the PK lead-in and in combination with BAY 1895344 will be compared with a non-parametric paired test, at a significance level at p < 0.05.
AUC and Cmax of BAY 1895344 | Up to 1 year post treatment
  PK of BAY 1895344 in combination with irinotecan and fluorouracil will be compared with historical controls in an exploratory fashion.
ATM status | Up to 1 year post treatment
  Will be assessed by immunohistochemistry (IHC) and PFS. The association between ATM and responses will be described, with a table outlining patients who achieved progressive disease, stable disease, partial or complete responses and whether they exhibited ATM expression by IHC or not.

OTHER OUTCOMES:
Incidence of adverse events | Up to 1 year post treatment
  Logistic regression and proportional hazards (Cox) regression will be used to assess the relationships between exposure and response and toxicity; exposure-response will be assessed within disease cohorts of sufficient size, while exposure-toxicity will pool all patients. All patients will be used for the E-R analyses. Advanced population PK methods may be employed at a later stage to assess the link between drug exposure and biological effects and efficacy.
Status of deoxyribonucleic acid damage repair (DDR) genes | Up to 1 year post treatment
  Assessed by whole exome sequencing and ribonucleic acid sequencing. The efficacy analyses will be repeated by DDR tumor mutation status, but these analyses will have limited sample sizes and will not be adequately powered for statistical comparisons.

CONTACTS AND LOCATIONS:
Overall Officials: Liza C Villaruz, Principal Investigator — University of Pittsburgh Cancer Institute LAO
Locations (10):
- United States (10):
  - City of Hope Comprehensive Cancer Center, Duarte, California
  - National Cancer Institute Developmental Therapeutics Clinic, Bethesda, Maryland
  - National Institutes of Health Clinical Center, Bethesda, Maryland
  - Siteman Cancer Center at Saint Peters Hospital, City of Saint Peters, Missouri
  - Siteman Cancer Center at West County Hospital, Creve Coeur, Missouri
  - Washington University School of Medicine, St Louis, Missouri
  - Siteman Cancer Center-South County, St Louis, Missouri
  - Siteman Cancer Center at Christian Hospital, St Louis, Missouri
  - NYP/Columbia University Medical Center/Herbert Irving Comprehensive Cancer Center, New York, New York
  - University of Pittsburgh Cancer Institute (UPCI), Pittsburgh, Pennsylvania

IPD SHARING:
Plan to Share IPD: Yes
NCI is committed to sharing data in accordance with NIH policy. For more details on how clinical trial data is shared, access the link to the NIH data sharing policy page.
URL: https://grants.nih.gov/policy/sharing.htm

REFERENCES:
- [Derived] Krishnamurthy A, Wang H, Rhee JC, Davar D, Moy RH, Ratner L, Christner SM, Holleran JL, Deppas J, Sclafani C, Schmitz JC, Gore S, Chu E, Bakkenist CJ, Beumer JH, Villaruz LC. Phase I trial of ATR inhibitor elimusertib with FOLFIRI in advanced or metastatic gastrointestinal malignancies (ETCTN 10406). Cancer Chemother Pharmacol. 2025 Jan 22;95(1):27. doi: 10.1007/s00280-024-04745-6. PMID 39841295